CLINICAL TRIAL: NCT04380870
Title: Describing Chinese Herbal Medicine Telehealth Care for Symptoms Related to Infectious Diseases Such as COVID-19: A Descriptive, Longitudinal, Pragmatic Cohort Study
Brief Title: Describing Chinese Herbal Medicine Telehealth Care for Symptoms Related to Infectious Diseases Such as COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Center for Integrated Care (Other)
Collaborators: University of Utah (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Katherine Taromina, Instructor, Supervisor, Center for Integrated Care
Other Study IDs: 01-04-20
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Coronavirus Infection
Keywords: COVID-19 symptoms; Chinese Herbal Medicine; Cough; Shortness of Breath; Fatigue; Epidemic; Infectious Disease; Dyspnea; Diarrhea; Myalgia; Nausea; Fever; Pneumonia
MeSH Terms: conditions — Coronavirus Infections; Cough; Dyspnea; Fatigue; Communicable Diseases; Diarrhea; Myalgia; Nausea; Fever; Pneumonia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese Herbal Medicine: Chinese Herbal Medicine for suspected COVID-19 symptoms.
  Interventions: Dietary Supplement: Chinese Herbal Medicine

INTERVENTIONS:
Dietary Supplement: Chinese Herbal Medicine — Chinese Herbal Medicine (CHM) has been used in the prevention and treatment of epidemic diseases dating back to the Han, Ming and Qing Dynasties and extending al the way through modern times. CHM formulas may contain plant elements of root, seed, back, stem or leaf in addition to minerals and other natural substances. All herbs dispensed in this trial will be from Spring Wind Herb Company.

SUMMARY:
The purpose of the study is to design and execute a prospective, longitudinal, descriptive cohort study in a pragmatic clinical practice for adults with symptoms that may be related to COVID-19.

DETAILED DESCRIPTION:
The purpose of this study is to design and execute a prospective, longitudinal, descriptive cohort study in a pragmatic clinical practice for adults with symptoms that may be related to COVID-19 infection who participate in Chinese herbal medicine (CHM) telehealth visits and take CHM. CHM includes over 400 medicinal substances and CHM formulas are individualized at each visit according to the patient's presentation. CHM has been used to treat cough, shortness of breath, and fatigue and mechanisms of action have been investigated for SARS and H1N1 influenza prevention and treatment by anti-inflammatory effects and antiviral activity. Yet, there is a gap in our understanding of the clinical application of CHM in a community sample of individuals experiencing symptoms that may be related to COVID-19. The investigators have no pragmatic clinic data about the use of CHM for coronaviruses.

Safe and effective treatment of symptoms associated with COVID-19 is a top international priority and research is needed to better understand if CHM is a safe intervention to treat symptoms. Further, dissemination of trustworthy CHM treatment approaches for this complex and emergent condition is needed within the CHM and scientific communities.

Aim 1: Conduct quantitative analyses of the collected data and disseminate findings to CHM clinicians and to the scientific community.

Case series will be reported bi-weekly to CHM clinicians via the SIEAM website including exposure, comorbidities, symptom change, concurrent medications, CHM prescriptions, adverse events and usability. Data will be analyzed at the study conclusion for presentation to the scientific community.

Aim 2: Conduct qualitative analyses of the collected data and disseminate findings to CHM clinicians and to the scientific community.

Chart notes reflecting clinicians' clinical reasoning will be content analyzed and posted bi-weekly on the SIEAM website. This will provide timely information for the CHM clinical community from highly experienced clinicians. Data will be analyzed at the study conclusion for presentation to the scientific community.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen year of age.
* Experienced one or more of the following symptoms in the last 28 days: cough, fever, shortness of breath, diarrhea, nausea, or abdominal pain OR am at high risk of exposure.
* Have a Primary Care Provider.

Exclusion Criteria:

* Breastfeeding, pregnant, or expect that I might be pregnant.
* Ineligible to receive a telehealth consult for any reason.
* Unable to communicate in English verbally, and in writing.
* Have an open legal case about my health.
* Taking anticoagulants, immunosuppressants, antiseizure medications, antipsychotic medications or am in active cancer treatment
* Taking medications with some risk of interaction with the herbal medicine. This will be determined at the time of the herbal consult by the clinic team.
* Discretion of the practitioner or screener.

Ages: 18 Years to 114 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-12-11 (Estimated); Study Completion 2025-05-11 (Estimated)

PRIMARY OUTCOMES:
Patient reported main complaint | 24 hours
  Patient reported change
Patient reported main complaint | 48 hours
  Patient reported change
Patient reported main complaint | 3 months
  Patient reported change
Patient reported main complaint | 12 months
  Patient reported change

SECONDARY OUTCOMES:
Conduct qualitative analyses of data | 24 hours
  Patient interview notes as written by clinicians.
Conduct qualitative analyses of data | 48 hours
  Patient interview notes as written by clinicians.
Conduct qualitative analyses of data | 3 months
  Patient interview notes as written by clinicians.
Conduct qualitative analyses of data | 12 months
  Patient interview notes as written by clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Taylor-Swanson, PhD, Principal Investigator — University of Utah; Lisa Conboy, DSc, Principal Investigator — Beth Israel Deaconness Medical Center, Harvard Medical School
Locations (1):
- Seattle Intstitute of East Asian Medicine, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Confidential, de-identified,demographic and health symptoms will be collected as part of this study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start with publication for a year.
Access Criteria: Site Principal Investigator to review written requests from HIPPA-trained investigators.

REFERENCES:
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Wong SH, Lui RN, Sung JJ. Covid-19 and the digestive system. J Gastroenterol Hepatol. 2020 May;35(5):744-748. doi: 10.1111/jgh.15047. Epub 2020 Apr 19. PMID 32215956
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] van Doremalen N, Bushmaker T, Morris DH, Holbrook MG, Gamble A, Williamson BN, Tamin A, Harcourt JL, Thornburg NJ, Gerber SI, Lloyd-Smith JO, de Wit E, Munster VJ. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med. 2020 Apr 16;382(16):1564-1567. doi: 10.1056/NEJMc2004973. Epub 2020 Mar 17. No abstract available. PMID 32182409
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Rodriguez-Morales AJ, Cardona-Ospina JA, Gutierrez-Ocampo E, Villamizar-Pena R, Holguin-Rivera Y, Escalera-Antezana JP, Alvarado-Arnez LE, Bonilla-Aldana DK, Franco-Paredes C, Henao-Martinez AF, Paniz-Mondolfi A, Lagos-Grisales GJ, Ramirez-Vallejo E, Suarez JA, Zambrano LI, Villamil-Gomez WE, Balbin-Ramon GJ, Rabaan AA, Harapan H, Dhama K, Nishiura H, Kataoka H, Ahmad T, Sah R; Latin American Network of Coronavirus Disease 2019-COVID-19 Research (LANCOVID-19). Electronic address: https://www.lancovid.org. Clinical, laboratory and imaging features of COVID-19: A systematic review and meta-analysis. Travel Med Infect Dis. 2020 Mar-Apr;34:101623. doi: 10.1016/j.tmaid.2020.101623. Epub 2020 Mar 13. PMID 32179124
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Yuen KS, Ye ZW, Fung SY, Chan CP, Jin DY. SARS-CoV-2 and COVID-19: The most important research questions. Cell Biosci. 2020 Mar 16;10:40. doi: 10.1186/s13578-020-00404-4. eCollection 2020. PMID 32190290
- [Background] Poston JT, Patel BK, Davis AM. Management of Critically Ill Adults With COVID-19. JAMA. 2020 May 12;323(18):1839-1841. doi: 10.1001/jama.2020.4914. No abstract available. PMID 32215647
- [Background] Sheahan TP, Sims AC, Graham RL, Menachery VD, Gralinski LE, Case JB, Leist SR, Pyrc K, Feng JY, Trantcheva I, Bannister R, Park Y, Babusis D, Clarke MO, Mackman RL, Spahn JE, Palmiotti CA, Siegel D, Ray AS, Cihlar T, Jordan R, Denison MR, Baric RS. Broad-spectrum antiviral GS-5734 inhibits both epidemic and zoonotic coronaviruses. Sci Transl Med. 2017 Jun 28;9(396):eaal3653. doi: 10.1126/scitranslmed.aal3653. PMID 28659436
- [Background] Colson P, Rolain JM, Raoult D. Chloroquine for the 2019 novel coronavirus SARS-CoV-2. Int J Antimicrob Agents. 2020 Mar;55(3):105923. doi: 10.1016/j.ijantimicag.2020.105923. Epub 2020 Feb 15. No abstract available. PMID 32070753
- [Background] Lai CC, Liu YH, Wang CY, Wang YH, Hsueh SC, Yen MY, Ko WC, Hsueh PR. Asymptomatic carrier state, acute respiratory disease, and pneumonia due to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2): Facts and myths. J Microbiol Immunol Infect. 2020 Jun;53(3):404-412. doi: 10.1016/j.jmii.2020.02.012. Epub 2020 Mar 4. PMID 32173241
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Chu CM, Cheng VC, Hung IF, Wong MM, Chan KH, Chan KS, Kao RY, Poon LL, Wong CL, Guan Y, Peiris JS, Yuen KY; HKU/UCH SARS Study Group. Role of lopinavir/ritonavir in the treatment of SARS: initial virological and clinical findings. Thorax. 2004 Mar;59(3):252-6. doi: 10.1136/thorax.2003.012658. PMID 14985565
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Atluri S, Manchikanti L, Hirsch JA. Expanded Umbilical Cord Mesenchymal Stem Cells (UC-MSCs) as a Therapeutic Strategy in Managing Critically Ill COVID-19 Patients: The Case for Compassionate Use. Pain Physician. 2020 Mar;23(2):E71-E83. PMID 32214286
- [Background] Conti P, Ronconi G, Caraffa A, Gallenga CE, Ross R, Frydas I, Kritas SK. Induction of pro-inflammatory cytokines (IL-1 and IL-6) and lung inflammation by Coronavirus-19 (COVI-19 or SARS-CoV-2): anti-inflammatory strategies. J Biol Regul Homeost Agents. 2020 March-April,;34(2):327-331. doi: 10.23812/CONTI-E. PMID 32171193
- [Background] Russell CD, Millar JE, Baillie JK. Clinical evidence does not support corticosteroid treatment for 2019-nCoV lung injury. Lancet. 2020 Feb 15;395(10223):473-475. doi: 10.1016/S0140-6736(20)30317-2. Epub 2020 Feb 7. No abstract available. PMID 32043983
- [Background] Ni L, Zhou L, Zhou M, Zhao J, Wang DW. Combination of western medicine and Chinese traditional patent medicine in treating a family case of COVID-19. Front Med. 2020 Apr;14(2):210-214. doi: 10.1007/s11684-020-0757-x. Epub 2020 Mar 13. PMID 32170559
- [Background] Chen MC, Lai JN, Chen PC, Wang JD. Concurrent Use of Conventional Drugs with Chinese Herbal Products in Taiwan: A Population-based Study. J Tradit Complement Med. 2013 Oct;3(4):256-62. doi: 10.4103/2225-4110.119734. PMID 24716186
- [Background] Runfeng L, Yunlong H, Jicheng H, Weiqi P, Qinhai M, Yongxia S, Chufang L, Jin Z, Zhenhua J, Haiming J, Kui Z, Shuxiang H, Jun D, Xiaobo L, Xiaotao H, Lin W, Nanshan Z, Zifeng Y. Lianhuaqingwen exerts anti-viral and anti-inflammatory activity against novel coronavirus (SARS-CoV-2). Pharmacol Res. 2020 Jun;156:104761. doi: 10.1016/j.phrs.2020.104761. Epub 2020 Mar 20. PMID 32205232
- [Background] Lau JT, Leung PC, Wong EL, Fong C, Cheng KF, Zhang SC, Lam CW, Wong V, Choy KM, Ko WM. The use of an herbal formula by hospital care workers during the severe acute respiratory syndrome epidemic in Hong Kong to prevent severe acute respiratory syndrome transmission, relieve influenza-related symptoms, and improve quality of life: a prospective cohort study. J Altern Complement Med. 2005 Feb;11(1):49-55. doi: 10.1089/acm.2005.11.49. PMID 15750363
- [Background] Luo H, Tang QL, Shang YX, Liang SB, Yang M, Robinson N, Liu JP. Can Chinese Medicine Be Used for Prevention of Corona Virus Disease 2019 (COVID-19)? A Review of Historical Classics, Research Evidence and Current Prevention Programs. Chin J Integr Med. 2020 Apr;26(4):243-250. doi: 10.1007/s11655-020-3192-6. Epub 2020 Feb 17. PMID 32065348
- [Background] Liu X, Zhang M, He L, Li Y. Chinese herbs combined with Western medicine for severe acute respiratory syndrome (SARS). Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD004882. doi: 10.1002/14651858.CD004882.pub3. PMID 23076910
- [Background] Duan ZP, Jia ZH, Zhang J, Liu S, Chen Y, Liang LC, Zhang CQ, Zhang Z, Sun Y, Zhang SQ, Wang YY, Wu YL. Natural herbal medicine Lianhuaqingwen capsule anti-influenza A (H1N1) trial: a randomized, double blind, positive controlled clinical trial. Chin Med J (Engl). 2011 Sep;124(18):2925-33. PMID 22040504
- [Background] Wang C, Cao B, Liu QQ, Zou ZQ, Liang ZA, Gu L, Dong JP, Liang LR, Li XW, Hu K, He XS, Sun YH, An Y, Yang T, Cao ZX, Guo YM, Wen XM, Wang YG, Liu YL, Jiang LD. Oseltamivir compared with the Chinese traditional therapy maxingshigan-yinqiaosan in the treatment of H1N1 influenza: a randomized trial. Ann Intern Med. 2011 Aug 16;155(4):217-25. doi: 10.7326/0003-4819-155-4-201108160-00005. PMID 21844547
- [Background] Coghlan ML, Maker G, Crighton E, Haile J, Murray DC, White NE, Byard RW, Bellgard MI, Mullaney I, Trengove R, Allcock RJ, Nash C, Hoban C, Jarrett K, Edwards R, Musgrave IF, Bunce M. Combined DNA, toxicological and heavy metal analyses provides an auditing toolkit to improve pharmacovigilance of traditional Chinese medicine (TCM). Sci Rep. 2015 Dec 10;5:17475. doi: 10.1038/srep17475. PMID 26658160
- [Background] Chen W, Liu B, Wang LQ, Ren J, Liu JP. Chinese patent medicines for the treatment of the common cold: a systematic review of randomized clinical trials. BMC Complement Altern Med. 2014 Jul 30;14:273. doi: 10.1186/1472-6882-14-273. PMID 25074623
- [Background] Yang Y, Islam MS, Wang J, Li Y, Chen X. Traditional Chinese Medicine in the Treatment of Patients Infected with 2019-New Coronavirus (SARS-CoV-2): A Review and Perspective. Int J Biol Sci. 2020 Mar 15;16(10):1708-1717. doi: 10.7150/ijbs.45538. eCollection 2020. PMID 32226288
- See also: Corona Resource Center — https://coronavirus.jhu.edu
- See also: WHO Coronavirus disease (COVID-19) situation dashboard — https://experience.arcgis.com/experience/685d0ace521648f8a5beeeee1b9125cd